CLINICAL TRIAL: NCT02542540
Title: Effects of a Physical Rehabilitation Program Using the Nintendo Wii on Children With Osteogenesis Imperfecta (OI) Is Nintendo Wii an Effective Intervention for Children With Osteogenesis Imperfecta
Brief Title: Effects of a Physical Rehabilitation Program Using the Nintendo Wii on Children With Osteogenesis Imperfecta (OI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty to include patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1201174
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-09

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; physical exercise training; Wii; muscular strength
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OI Children training with Nintendo Wii console (Experimental): Training for 3 months using the Nintendo Wii console on physical capacity in a group of children with Osteogenesis Imperfecta
  Interventions: Other: Training with Nintendo Wii console
- Children with OI without training (No Intervention): No training

INTERVENTIONS:
Other: Training with Nintendo Wii console — Children with OI and draining for 3 months using Nintendo Wii console
  Arms: OI Children training with Nintendo Wii console

SUMMARY:
Children with osteogenesis imperfecta are described as extremely sedentary and therefore fatigable, which strongly impacts their daily activities. The physical rehabilitation of these children is a fundamental aspect of treatment.

It has been shown that playing Wii console causes the same increase in energy expenditure than practicing moderate exercise, while ensuring user safety. This type of physical exercise with this type of fun game console might have a role in the treatment of OI children on the physical side but also on the psychological side.

ELIGIBILITY:
Inclusion Criteria:

* - Children affiliated to a social security scheme
* Children diagnosed OI by a competent physician of one of the French specialist centers;
* OI children type 1 or type 4;
* Stable OI (far from a fractional episode of at least two months);
* Children without regular activity on the Nintendo Wii console or other interactive console;
* Boy or Girl> 6 to 18 years
* Parents or person having parental authority affiliated to a social security scheme
* Parents or person having parental authority who signed the consent form for the study.

Exclusion Criteria:

* - Children who can not walk;
* Children with severe OI other than type 1 or type 4;
* Fracture during the last two months;
* Surgical intervention within the last 8 months;
* Inability to understand and follow the protocol;
* Participation in another clinical study;
* Children, parents or holder of parental authority refusing the written consent.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in physical capacity | from baseline to 3 months
  Compare the change in physical capacity between training group of children with OI and control group of children with OI. The physical capacity is measured by maximal oxygen consumption VO2 max (ml/min/kg) measured during incremental exercise on cycle ergometer

SECONDARY OUTCOMES:
Change in physical capacity | From baseline to 9 months
  Compare the change in physical capacity between training group of children with OI and control group of children with OI. The physical capacity is measured by maximal oxygen consumption VO2 max (ml/min/kg) measured during incremental exercise on cycle ergometer
Compare physical inactivity between training group and control group | Month 3
  Physical inactivity will be assessed by the Physical Activity Questionnaire (Q-APS)
Compare physical inactivity between training group and control group | Month 9
  Physical inactivity will be assessed by the Physical Activity Questionnaire (Q-APS)
Compare functional benefit between training group and control group | Month 3
  The functional benefit will be evaluated by the Functional Independence Measure (FIM)
Compare functional benefit between training group and control group | Month 9
  The functional benefit will be evaluated by the Functional Independence Measure (FIM)
Compare body fat between training group and control group | Month 3
  Body fat composition will be determined by skinfold measurements
Compare body fat between training group and control group | Month 9
  Body fat composition will be determined by skinfold measurements
Compare quality of life between training group and control group | Month 3
  The quality of life will be determined the Index Questionnaire Reintegration to Normal Life (IRVN)
Compare quality of life between training group and control group | Month 9
  The quality of life will be determined the Index Questionnaire Reintegration to Normal Life (IRVN)
Compare muscle strength between training group and control group | Month 3
  The muscle strength is a composite outcome. It will be assessed by:
  * The grip strength (force applied by the hand)
  * The maximal quadriceps muscle strength will be measured using an isokinetic dynamometer "Contrex"
Compare muscle strength between training group and control group | Month 9
  The muscle strength is a composite outcome. It will be assessed by:
  * The grip strength (force applied by the hand)
  * The maximal quadriceps muscle strength will be measured using an isokinetic dynamometer "Contrex"
Compare endurance of lower limbs between training group and control group | Month 3
  The endurance of the lower limbs will be measured by EMG analysis on incremental torque repetitive exercise
Compare endurance of lower limbs between training group and control group | Month 9
  The endurance of the lower limbs will be measured by EMG analysis on incremental torque repetitive exercise
Compare Energy expenditure of lower limbs between training group and control group | Month 3
  Energy expenditure is a composite outcome. It will be measured by collecting the respiratory exchange and heart rate during endurance, tennis and boxing games using the Nintendo WII
Compare Energy expenditure of lower limbs between training group and control group | Month 9
  Energy expenditure is a composite outcome. It will be measured by collecting the respiratory exchange and heart rate during endurance, tennis and boxing games using the Nintendo WII
Training tolerance | Baseline from 9 months
  Reentrainment tolerance is a composite outcome. It will be assessed by :
  * collecting any events related to WII training or any events related to everyday life (fractures, pain,etc.)
  * dropout rate study report

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gautheron, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France